CLINICAL TRIAL: NCT05792969
Title: Public Health Impact of Unilateral Spatial Neglect
Acronym: IMPAssNEGLECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 25C123
Record Dates: First submitted 2023-03-03; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Spatial Neglect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients with USN and their caregivers
  Interventions: Behavioral: Functional measures and public health outcomes
- Stroke patients without USN and their caregivers
  Interventions: Behavioral: Functional measures and public health outcomes

INTERVENTIONS:
Behavioral: Functional measures and public health outcomes — Questionnaires:
  * Activities of daily living - ADL
  * Barthel Index
  * Instrumental activities of daily living- IADL
  * Health Related Quality of Life - EQ-5D-5L
  * Geriatric Depression Scale (GDS)
  * State-Trait Anxiety Inventory - STAI-Y)
  * Caregiver Burden Inventory questionnaire (CBI)

SUMMARY:
This multi-center project aims to quantify the socio-medical costs associated with Unilateral Spatial Neglect (USN) resulting from acquired brain injury (stroke) and to measure the effects of USN rehabilitation on functional autonomy, quality of life and psychological well-being of patients affected by this syndrome, considering the repercussions on a psychological level and on the quality of life of caregivers.

To this end, the experimenters will administer to right brain-injured patients - with (Experimental Group) or without (Control Group) USN - who undertook a rehabilitation process, a series of questionnaires: Activities of daily living (ADL), Barthel Index; Instrumental activities of daily living scale (I-ADL:), the Health Related Quality of Life questionnaire (EQ-5D-5L), the Geriatric Depression Scale (GDS), and the State-Trait Anxiety Inventory (STAI-Y). The aforementioned tests will be administered before the start of the rehabilitation (baseline) and after one month, 3, 6 and 12 months after the end of the rehabilitation. The impact of USN and its treatment on the psycho-physical well-being of the caregiver will be measured through the Caregiver Burden Inventory questionnaire, which will be administered with the same timing (baseline, 1-3-6-12 months after rehabilitation). The costs of USN will be surveyed through an ad-hoc questionnaire, which includes a version intended for patients and one for caregivers, in order to identify the resources consumed due to the disease and the expenses taken during the observation period, to be estimated subsequently in monetary terms (€).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* right brain injury due to stroke (of ischemic or hemorrhagic origin);
* Disease duration ≥ 10 days;
* Participation to a rehabilitation program;

For stroke patients with USN:

- clinical diagnosis of USN, placed by the specialist of reference, on the basis of clinical indicators and the results obtained by the patient in the routine neuropsychological evaluation (by means of a battery of standardized psychometric tests calibrated in the Italian population).

Exclusion Criteria:

* Other brain disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients with and without USN and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Activities of Daily Living scale (ADL) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  To evaluate the degree of patients' functional independence in everyday life
Change in the Instrumental Activities of Daily Living scale (I-ADL) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  To evaluate the degree of patients' functional independence instrumental activities, including, e.g., cleaning, cooking, and managing finances.
Change in the Health-Related Quality of Life (EQ-5D-5L) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  A brief scale assessing patient's health-related quality of life
Change in the Geriatric Depression Scale (GDS) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  A scale assessing patients' depressive symptoms
Change in the State-Trait Anxiety Inventory (STAI-Y) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  A scale assessing patients' anxiety symptoms
Change in the Caregiver Burden Inventory questionnaire (CBI) | At baseline (at the beginning of the treatment) and after 1, 3, 6, and 12 months after the end of the treatment
  A scale that assess caregivers' physical and psychological burden
Financial impact of USN | 1 month after the end of the treatment
  A questionnaire about health-related costs associated to the disease (e.g., heath examinations, medicines, sick leaves)
Financial impact of USN | 3 months after the end of the treatment
  A questionnaire about health-related costs associated to the disease (e.g., heath examinations, medicines, sick leaves)
Financial impact of USN | 6 months after the end of the treatment
  A questionnaire about health-related costs associated to the disease (e.g., heath examinations, medicines, sick leaves)
Financial impact of USN | 12 months after the end of the treatment
  A questionnaire about health-related costs associated to the disease (e.g., heath examinations, medicines, sick leaves)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy